CLINICAL TRIAL: NCT03617679
Title: A Phase II, Randomized, Double-Blind Study of the Use of Rucaparib vs. Placebo Maintenance Therapy in Metastatic and Recurrent Endometrial Cancer
Brief Title: Rucaparib vs Placebo Maintenance Therapy in Metastatic and Recurrent Endometrial Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Clovis Oncology, Inc. (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18-0567.cc; P30CA046934 (NIH)
Record Dates: First submitted 2018-07-17; First posted 2018-08-06 (Actual); Results first posted 2024-07-01 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Endometrial Cancer
Keywords: Rucaparib; Placebo; Randomized; Double Blind; Stage III/IV
MeSH Terms: conditions — Endometrial Neoplasms | interventions — rucaparib

STUDY DESIGN:
Intervention Model Description: Active ingredient vs placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Ingredient (Active Comparator): 1:1 Randomization. Participants in this arm receive the active ingredient medication.
  Interventions: Drug: Rucaparib
- Placebo (Placebo Comparator): 1:1 Randomization. Participants in this arm receive the placebo medication. (Placebos do not contain active ingredients).
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Rucaparib — Participants allocated to the active ingredient arm will receive Rucaparib twice daily, 600mg, to be take by mouth. Patients will take the medication continuously over a 28 day cycle, until disease progression or other indication of discontinuation. Medication should be taken around the same time every day, with 8 or more ounces of water.
  Arms: Active Ingredient
Drug: Placebo Oral Tablet — Participants allocated to the placebo arm will receive a placebo tablet (that looks identical to the active ingredient tablet) twice daily, 600mg, to be take by mouth. Patients will take the medication continuously over a 28 day cycle, until disease progression or other indication of discontinuation. Tablet should be taken around the same time every day, with 8 or more ounces of water.
  Arms: Placebo

SUMMARY:
This study seeks to determine the effectiveness of Rucaparib as maintenance therapy for metastatic and recurrent endometrial cancer, after 1-2 prior lines of therapy.

DETAILED DESCRIPTION:
This is a phase II clinical trial, that administers a maintenance treatment after first line chemotherapy is complete. It is designed to have a 1:1 randomization technique. Half the participants who enter the study will receive the active ingredient, Rucaparib, while the other half will receive a placebo. Treatment will be until progression with follow up until death.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be a female aged 18-89.
4. Patients with a primary Stage III/IV or recurrent endometrial cancer.
5. Patients have received at least one prior chemotherapy regimen and no more than two prior cytotoxic regimens (including hormonal therapy).
6. Primary chemotherapy regimen must have consisted of at least 4 completed cycles and no more than 8 completed cycles.
7. Previous cytotoxic regimen at least 4 weeks before initiation and no more than 8 weeks from initiation after last dose of previous therapy.
8. Patients who receive radiation to the whole pelvis or at least 50% of the spine must complete radiation therapy and have at least 4 weeks' time elapse prior to initiation of drug.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2.
10. Absolute neutrophil count (ANC) > or = 1500 cells/microliters
11. Platelet count > 100,000 microliters
12. Hemoglobin > or = 9.0 g/dL
13. Serum albumin > or = 2.5 g/dL
14. Total bilirubin ≤ 1.5 x ULN (uppler limit of normal)
15. AST and ALT ≤ 3.0 x ULN
16. Serum Creatinine ≤ 1.5x ULN

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Inability to comply with study and follow-up procedures
2. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within the past 3 months, unstable arrhythmias, or unstable angina
3. Known clinically significant liver disease defined as AST and ALT > 3.0 x ULN and/or Total bilirubin > or = 1.5 x ULN, or documented history of active viral, alcoholic, or other hepatitis, cirrhosis, and inherited liver disease
4. Participation in investigational clinical trial within last 30 days
5. History of significant chronic disease including HIV/AIDS or hepatitis C
6. Inability to provide informed consent
7. Known central nervous system (CNS) malignancy or CNS metastases
8. Patients with previous malignancy, other than endometrial, within the past 2 years from cycle 1, day 1, with the exception of those with negligible risk of metastasis or death, such as adequately controlled basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the breast.
9. History of stroke or transient ischemic attack (TIA) within 3 months prior to cycle 1 day 1(C1D1)
10. Women with prognosis for survival less than 6 months
11. Patients who have progressed or have stable disease (SD) through most recent chemotherapy regimen
12. Patients deemed otherwise clinically unfit for clinical trial per Investigator's discretion
13. Patients with duodenal stent or other GI disorder/defect that would interfere with absorption of oral medication
14. Female patients who maintain fertility potential and refuse to comply to use contraception and be followed for pregnancy by pregnancy testing
15. Minor surgical procedure < or = 14 days or major surgeries < or = 28 days prior to first dose of treatment

Ages: 18 Years to 89 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 79 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2025-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Corr, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Corr BR, Haggerty A, Gysler SM, Taylor S, Behbakht K, Alldredge J, Lefkowits C, Brubaker LW, Bouts C, Babayan LM, Martin LP, Costello J, Bitler BG, Hu J, Guntupalli SR. A phase II, randomized, double-blind study of the use of rucaparib vs. placebo maintenance therapy in metastatic and recurrent endometrial cancer. Gynecol Oncol. 2025 Sep;200:58-67. doi: 10.1016/j.ygyno.2025.07.008. Epub 2025 Jul 22. PMID 40700852

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Ingredient | Placebo
Started | 39 | 40
Completed | 39 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Ingredient | Placebo | Total
Number analyzed (Participants) | 39 | 40 | 79
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 21 | 23 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [61 to 72] | 67 [58 to 71] | 66 [59 to 71.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 40 | 79
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 35 | 38 | 73
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 3 | 7
  White | 33 | 34 | 67
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 40 | 79

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression free survival is defined as cycle 1 day 1 (C1D1) till the time of progression as determined by RECIST 1.1 criteria or death.
Time Frame: Up to 48 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Active Ingredient | Placebo
Number analyzed (Participants) | 39 | 40
months | 28.1 [12.8 to NA] — insufficient number of participants with events | 8.7 [5.4 to 16.7]

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as cycle 1 day 1 (C1D1) till the time of death.
Time Frame: Up to 48 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Active Ingredient | Placebo
Number analyzed (Participants) | 39 | 40
months | NA [34.8 to NA] — insufficient number of participants with events | 28.4 [19.0 to NA] — insufficient number of participants with events

3. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Safety and tolerability analysis of Rucaparib will be summarized by dose and severity as assessed by the Common Toxicity Criteria for Adverse Events (CTCAE) version 5 and relationship to study drug.
Time Frame: Up to 48 months.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Ingredient | Placebo
Number analyzed (Participants) | 39 | 40
Participants | 37 | 27

ADVERSE EVENTS:
Time Frame: 4 years and 8 months.
Arm/Group | Active Ingredient | Placebo
All-Cause Mortality (participants affected / at risk) | 1/39 | 1/40
Serious Adverse Events (participants affected / at risk) | 3/39 | 1/40
Other Adverse Events (participants affected / at risk) | 37/39 | 27/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Ingredient (N=39) | Placebo (N=40)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
elevated ALT/AST (Investigations) | 0 (0) | 1 (1)
neutropenia (Investigations) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Ingredient (N=39) | Placebo (N=40)
nausea (Gastrointestinal disorders) | 23 (23) | 9 (9)
fatigue (General disorders) | 24 (24) | 11 (11)
anemia (Blood and lymphatic system disorders) | 26 (26) | 8 (8)
thrombocytopenia (Investigations) | 15 (15) | 5 (5)
elevated ALT/AST (Investigations) | 13 (13) | 0 (0)
Dysgeusia (Nervous system disorders) | 8 (8) | 0 (0)
neutropenia (Investigations) | 9 (9) | 7 (7)
elevated alkaline phosphatase (Investigations) | 4 (4) | 1 (1)
dizziness (Nervous system disorders) | 4 (4) | 0 (0)
anorexia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
diarrhea (Gastrointestinal disorders) | 2 (2) | 4 (4)
dry mouth (Gastrointestinal disorders) | 2 (2) | 2 (2)
rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
hot flashes (Vascular disorders) | 2 (2) | 0 (0)
elevated creatinine (Investigations) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT03617679/Prot_SAP_000.pdf